CLINICAL TRIAL: NCT02894203
Title: Psychological and Biological Effects of Intensive Mindfulness Meditation on Offenders With Dangerous and Severe Personality Disorder: A Randomised Controlled Trial
Brief Title: Psychobiological Effects of Meditation on Offenders With Psychopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Coventry University (Other)
Collaborators: Donders Centre for Cognitive Neuroimaging (Other)
Responsible Party: Principal Investigator, Ivana Buric, MA, Doctoral candidate, Coventry University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 13274-24
Record Dates: First submitted 2016-08-30; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Mindfulness; Yoga
MeSH Terms: interventions — Mindfulness; Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mindfulness (Experimental)
  Interventions: Behavioral: Mindfulness
- Hatha Yoga (Active Comparator)
  Interventions: Behavioral: Yoga
- Wait-list (No Intervention)

INTERVENTIONS:
Behavioral: Mindfulness
  Arms: Mindfulness
Behavioral: Yoga
  Arms: Hatha Yoga

SUMMARY:
The investigators aim to explore the psychobiological effects of a 5-day meditation intervention on offenders within dangerous and severe personality disorders (DSPD) unit at HMP Whitemoor. DSPD unit accommodates offenders with psychopathy or with two or more personality disorders. DPSD unit provides them with a 5-year rehabilitation programme that consists of group and individual therapy and aims to improve their self-regulation.

This project includes a total of 60 participants and has two major methodological innovations. First, it will include yoga as an active control group that will be matched to the meditation intervention (which means it will have the same length and the same social components) and a passive control group that will be following their usual regimen. Thus, the effects of meditation will be contrasted with another type of intervention and with not receiving any intervention.

The second methodological innovation is the combination of psychological and biological measures. Psychological measures include questionnaires (emotion regulation, mindfulness, stress) and cognitive measures (attention,empathy,behavioural control). Biological measures include EEG to measure brain activity related to empathy; gene expression and protein interlukin-6 to measure changes in immune system; and stress related hormone cortisol. The investigators also aim to determine to whom does meditation benefit the most by exploring how initial expectations of meditation, personality, mood and previous life adversity predict outcomes of meditation or yoga. The data will be collected at three time points: at baseline, immediately after and 10 weeks after the 5-day intervention.

The investigators expect that meditation and yoga will similarly improve mental and physical health. If this hypothesis are confirmed, these results will extend previous findings on the benefits of meditation and yoga to vulnerable populations, and would provide a cost-effective addition to prisoner rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Male offenders with dangerous and severe personality disorder aged 18-65 who will remain in the prison until at least February 2017.

Exclusion Criteria:

* Major psychiatric or neurological disorders, previous meditation or yoga experience, unable to follow instructions in English,

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline emotional regulation | Before the intervention, up to 2 weeks after the intervention and at 10-18 week follow-up
  Difficulties in Emotion Regulation Scale
Change from baseline attention | Before the intervention, up to 2 weeks after the intervention and at 10-18 week follow-up
  Attention Network Task
Change from baseline self-awareness | Before the intervention, up to 2 weeks after the intervention and at 10-18 week follow-up
  Mindful Attention Awareness Scale
Change from baseline inflammatory gene expression | Before the intervention and on the final day of the intervention

SECONDARY OUTCOMES:
Change from baseline social learning | Before the intervention, up to 2 weeks after the intervention and at 10-18 week follow-up
  Social Learning Task (Diaconescu et al., 2014)
Change from baseline risk-taking | Before the intervention, up to 2 weeks after the intervention and at 10-18 week follow-up
  Risk-taking Task (Tymula et al., 2012)
Change from baseline empathy | Before the intervention, up to 2 weeks after the intervention and at 10-18 week follow-up
  Self-assessment Manikin (Seara & Cardoso, 2012).
Change from baseline stress | Before the intervention, up to 2 weeks after the intervention and at 10-18 week follow-up
  Perceived Stress Scale
Change from baseline affective states | Before the intervention, up to 2 weeks after the intervention and at 10-18 week follow-up
  Profile of Mood States

IPD SHARING:
Plan to Share IPD: Undecided